CLINICAL TRIAL: NCT03296462
Title: Physiotherapy for Stress Urinary Incontinence: Feasibility Study for a Randomized Controlled Trial of Hip External Rotation Exercise Training Versus Pelvic Floor Muscle Exercise Training
Brief Title: Hip External Rotation Physical Therapy Trial
Acronym: HER-Physio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Physiotherapy Alberta - College + Association (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00066652
Record Dates: First submitted 2017-09-18; First posted 2017-09-28 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Urinary Incontinence, Stress
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Patient and research assistant are blind to next allocation. Outcome assessors (physiotherapist and exercise physiologist) and one investigator are blinded to group of allocation. Statistician will be masked to group of allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hip external rotation exercise (alone) (Experimental): Standardised hip external rotation exercise training - over 12 week period
  Interventions: Other: Hip external rotation exercise
- Hip external rotation + PFM exercises (Experimental): Standardised hip external rotation plus pelvic floor muscle exercises - over 12 week period
  Interventions: Other: Hip external rotation exercise; Other: Pelvic floor muscle exercise
- pelvic floor muscle exercises (alone) (Active Comparator): Standardised pelvic floor muscle exercises - over 12 week period (usual care)
  Interventions: Other: Pelvic floor muscle exercise

INTERVENTIONS:
Other: Hip external rotation exercise — Standardised HER exercise training by physiotherapist (plus video recording of exercises)
  Arms: Hip external rotation + PFM exercises; Hip external rotation exercise (alone)
Other: Pelvic floor muscle exercise — Standardised PFM exercise training by physiotherapist (plus video recording of exercises)
  Arms: Hip external rotation + PFM exercises; pelvic floor muscle exercises (alone)

SUMMARY:
This RCT is a feasibility study to evaluate the Lois Hole Hospital for Women's Urogynecology Clinic's ability to recruit and randomize SUI patients to the proposed RCT, and to test the study procedures and follow-up schedule for participants.

The study interventions used in the feasibility study will be training of (1) Hip Extension Rotation (HER) exercises alone, (2) HER exercises in combination with Pelvic Floor Muscle (PFM) exercises, or (3) PFM exercises alone (control/usual care) in the treatment of SUI.

DETAILED DESCRIPTION:
Background: Hip External Rotation (HER) exercises are being adopted into physiotherapy practice for the treatment of stress urinary incontinence (SUI) despite little evidence compared to the proven effective standard of care treatment, pelvic floor muscle (PFM) exercises. A randomised clinical trial (RCT) is needed to determine whether HER exercise alone or in combination with PFM is more or less effective than PFM exercises alone.

Objective: Before designing an RCT, a feasibility study is needed to evaluate the Lois Hole Hospital for Women's Urogynecology Clinic's ability to recruit and randomize SUI patients to the proposed RCT, and to test the study procedures and follow-up schedule for participants.

Interventions: The interventions used in the feasibility study will be training of (1) HER exercises alone, (2) HER exercises in combination with PFM exercises, or (3) PFM exercises alone (control/usual care) in the treatment of SUI.

Study design: RCT in which participants are randomly allocated 1:1:1 to each intervention.

Outcome Measures: Feasibility outcomes will pertain to recruitment, adherence to training, appropriateness of outcome measures and completion rates. The design of the proposed RCT will be based on these feasibility outcomes.

Outcome measures for the proposed RCT will include pelvic floor muscle strength, external hip rotator muscle strength, diary-reported urinary incontinence, incontinence related quality of life, and (to test patient mobility) six minute walk test and timed up and go test.

Sample size: The proposed sample size is 30 participants. Duration of study: After recruitment, each woman will undergo 12 weeks of training, with the first outcome measure at the end of that period, and a further follow up at 24 weeks from recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Stress urinary incontinence
* Attending Lois Hole Hospital for Women Urogynecology Clinic
* Referred for physiotherapy for stress urinary incontinence
* Able to toilet independently
* Able to undertake hip rotation exercises
* Able to speak and read English

Exclusion Criteria:

* Urge urinary incontinence
* Using a pessary
* Neurological or cognitive impairment
* Using other treatment for incontinence
* Unable to complete study forms
* Unable to understand educational instruction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Feasibility: achieve recruitment of 30 women over 12 months | 12 months
  Is recruitment feasible? "Feasibility" is defined as achieving recruitment target of 30 recruits within 12 months
Feasibility: achieve follow-up for 60% of recruits over 12 months | 12 months
  Is follow-up complete for 60% of recruits?

SECONDARY OUTCOMES:
Pelvic floor muscle strength | 12 & 24 weeks
  Strength will be measured using Peritron perineometer
External hip rotator muscle strength | 12 & 24 weeks
  Strength will be measured using Microfit ET3
Diary-reported urinary incontinence | 12 & 24 weeks
  3-day bladder diary to record amount and reason for leakage
Incontinence-related quality of life (distress) | 12 & 24 weeks
  UDI-6 questionnaire (measure of distress caused by incontinence, 0 minimum to 100 maximum)
Incontinence-related quality of life (impact) | 12 & 24 weeks
  IIQ-7 questionnaire (measure of impact of incontinence, 0 minimum to 100 maximum)
Patient mobility (walking) | 12 & 24 weeks
  Six minute walk test - distance walked (metres)
Patient mobility | 12 & 24 weeks
  "timed up and go" test - time in sconds

CONTACTS AND LOCATIONS:
Overall Officials: Sue Ross, PhD, Study Director — University of Alberta
Locations (1):
- Lois Hole Hospital for Women, Royal Alexandra Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322